CLINICAL TRIAL: NCT00315068
Title: The Value of Amino-Terminal Brain Natriuretic Peptide and C-Reactive Protein Serum Levels for Predicting Recurrence of Atrial Fibrillation and/or Atrial Flutter After Radiofrequency Catheter Ablation
Brief Title: Usefulness of Markers to Predict Recurrence of Atrial Fibrillation After Radiofrequency Catheter Ablation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Geneva (Other)
Other Study IDs: PRD-03-I-03
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Atrial Fibrillation
Keywords: arrythmia; atrial fibrillation; proteins
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Catheter ablation using radiofrequency is a new therapeutic tool to treat atrial fibrillation with a higher success rate than medical therapy (80% versus less than 50% respectively). Because of the length of the intervention and of the risk of complications of the procedure, it would be important to determine success rate before the intervention. The information gained from this study will in all probability improve our estimation of the chances of a successful intervention and may enable us to take necessary therapeutic measures in case of an elevated risk of recurrence.

Multiple studies suggest that the 2 markers in this study could provide information of this nature, however, their utility in the radiofrequency catheter ablation treatment of atrial fibrillation has never been demonstrated.

DETAILED DESCRIPTION:
Catheter ablation of atrial fibrillation is a recent therapeutic tool to treat atrial fibrillation. The success rate of eliminating atrial fibrillation by radiofrequency catheter ablation is 80 %, after one or sometimes two procedures, against 20-50 % with drug treatment.

This intervention may be complicated by : hematoma at the puncture site - 1 % incidence; thromboembolic events < 1 % incidence; cardiac perforation with tamponade < 1 %, pulmonary vein stenosis 2 % incidence.

The aim of this study is to evaluate blood tests of biological products (NT-proBNP and CRP) as markers of prognosis and success after radiofrequency catheter ablation for atrial fibrillation.

Previous studies demonstrated the prognostic value of NT-proBNP and CRP in the recurrence of atrial fibrillation after electrical cardioversion. However the prognostic value of these biomarkers was never demonstrated in the setting of radiofrequency catheter ablation of atrial fibrillation.

This is an observation study including 180 patients with the indication of catheter ablation for atrial fibrillation. Confounding factors of increased NT-proBNP will be assessed with echocardiographic imaging.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation
* indication for catheter ablation of atrial fibrillation

Exclusion Criteria:

* significant valvulopathy
* previous catheter ablation for atrial fibrillation or atrial flutter
* left ventricular ejection fraction < 30%
* Severe heart failure (NYHA IV)
* Severe enlargement of left atrium (> 55mm)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2004-04; Study Completion 2007-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Frederic Keller, MD, Principal Investigator — Cardiology Division University Hospital
Locations (1):
- Cardiology Division University Hospital, Geneva, Canton of Geneva, Switzerland